CLINICAL TRIAL: NCT04527471
Title: A Single-center, Pilot, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Ensifentrine in the Recovery of Hospitalized Patients With COVID-19
Brief Title: Pilot Study of Ensifentrine or Placebo Delivered Via pMDI in Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma Inc (Industry)
Responsible Party: Sponsor
Organization: Verona Pharma plc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPL554-COV-201
Record Dates: First submitted 2020-08-06; First posted 2020-08-26 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus Infection; Covid-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ensifentrine + Standard of Care (Active Comparator): 30 subjects randomized to receive blinded, inhaled ensifentrine in addition to standard of care treatment for COVID-19 infection
  Interventions: Drug: Ensifentrine Dose 1
- Placebo + Standard of Care (Placebo Comparator): 15 subjects randomized to receive blinded, inhaled placebo in addition to standard of care treatment for COVID-19 infection
  Interventions: Drug: Placebo pMDI

INTERVENTIONS:
Drug: Ensifentrine Dose 1 — Study drug delivered twice daily via pMDI
  Arms: Ensifentrine + Standard of Care
Drug: Placebo pMDI — Placebo delivered twice daily via pMDI
  Arms: Placebo + Standard of Care

SUMMARY:
This pilot study is being performed to assess the efficacy and safety of inhaled ensifentrine delivered via pMDI compared with a matching placebo in conjunction with standard of care treatments on recovery in patients hospitalized due to COVID-19 infection.

DETAILED DESCRIPTION:
Expploratory endpoint, pilot study, not statistically powered

go to protocol

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent indicating that they understand the purpose of the study and study procedures and agree to comply with the requirements and restrictions listed in the informed consent form and in this protocol.
* Patient must be at least 18 years of age and less than or equal to 80 years of age at the time of informed consent.
* Males are eligible to participate or females of non-childbearing potential or WOCBP who have a negative pregnancy test at screening are eligible to participate. WOCBP and female partners of male participants agree to either abstinence or use at least one primary form of highly effective contraception not including hormonal contraception from the time of screening through Day 60 following the first dose of study medication.
* Clinical status consistent with 3, 4 or 5 on the Ordinal scale: Hospitalized, not requiring supplemental oxygen; Hospitalized, requiring any supplemental oxygen; Hospitalized, requiring non-invasive ventilation or use of high flow oxygen devices.
* Admission to hospital AND have a confirmed diagnosis of severe acute respiratory syndrome coronavirus (SARS-COV-2) infection confirmed by polymerase chain reaction (PCR) test AND displays at least one of the following: Respiratory rate > 24 breaths per minute; new cough; new atypical chest pain; new dyspnea; oxygen saturation < 97% at rest; chest x-ray with new changes consistent with COVID-related airspace disease.
* Capable of complying with all study restrictions and procedures including ability to use the pMDI correctly.

Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment for COVID-19, unless related to an expanded access program as part of Standard of Care at screening or during study.
* Evidence of multiorgan failure.
* Requiring mechanical ventilation at screening.
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN) at screening.
* Creatinine clearance < 30 mL/min at screening.
* Pregnancy or lactation at screening.
* Allergy or other contraindication or one of ensifentrine.
* In the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
* Use of prohibited medications (theophylline, PDE4 inhibitors [e.g. roflumilast, apremilast, crisaborole] within 48 hours of screening or during study)
* Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Verona Pharma will not be sharing individual deidentified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 patients hospitalized with COVID-19 enrolled and randomized.
Pre-assignment Details: 45 patients randomized to receive either RPL554 2mg via pMDI BID or placebo via pMDI BID in addition to standard of care treatment for COVID-19 disease until discharged or Day 29, whichever was first.
Period: Overall Study
Arm/Group | Ensifentrine + Standard of Care | Placebo + Standard of Care
Started | 30 | 15
Hospitalized up to 7 Days | 24 | 12
Hospitalized for > 7 Days | 6 | 3
Completed (Through Day 60 Follow-up) | 28 | 15
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ensifentrine + Standard of Care | Placebo + Standard of Care | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (13.3) | 51.5 (14.7) | 56.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 14 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 21 | 8 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 15 | 45
COVID-19 Disease Severity (Moderate) [Count of Participants; unit: Participants] | 30 | 15 | 45
Smoking Status (Previous) [Count of Participants; unit: Participants] | 7 | 1 | 8
Supplemental Oxygen Use (Yes) [Count of Participants; unit: Participants] | 30 | 14 | 44
2 or more Co-Morbidities [Count of Participants; unit: Participants] | 16 | 4 | 20
Systolic Blood Pressure [Median (Full Range); unit: mmHg] | 145 [86 to 174] | 124 [96 to 170] | 138 [86 to 174]
Smoking Status (Current) [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Recovery
Description: Recovery = first day on which subject satisfies one of the following categories: not hospitalized, no limitations of activities; or not hospitalized, limitation of activities, home oxygen requirement, or both.
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Ensifentrine + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 30 | 15
Participants | 29 | 15
Statistical Analysis 1: Comparison: Ensifentrine + Standard of Care vs Placebo + Standard of Care; Test type: Other; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: Over 60 days
Arm/Group | Ensifentrine + Standard of Care | Placebo + Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/15
Other Adverse Events (participants affected / at risk) | 5/30 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensifentrine + Standard of Care (N=30) | Placebo + Standard of Care (N=15)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensifentrine + Standard of Care (N=30) | Placebo + Standard of Care (N=15)
Sinus bradycardia and Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This was an un-powered pilot study of ensifentrine pMDI in patients hospitalized for moderate COVID-19 infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT04527471/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04527471/SAP_001.pdf